CLINICAL TRIAL: NCT04613050
Title: Effect of Respiratory Versus Aerobic Training on Respiratory and Immunity Efficiency in Recovered COVID- 19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAHA2020
Record Dates: First submitted 2020-10-30; First posted 2020-11-03 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Covid 19 Infection
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Respiratory Training Group) (Active Comparator): It will include 30 patients of both sexes, recovered from COVID-19 infection. In addition to medical drugs, they will receive respiratory training for 6 weeks.
  Interventions: Other: Respiratory Training
- Group B : (Aerobic Training Group) (Active Comparator): It will include 30 patients of both sexes, recovered from COVID-19 infection. In addition to medical drugs, they will receive aerobic training for 6 weeks
  Interventions: Other: Aerobic training
- Group C : (control group) (No Intervention): It will include 20 patients of both sexes, recovered from COVID-19 infection on medical drugs only will receive no exercise as control group.

INTERVENTIONS:
Other: Respiratory Training — Respiratory training in form of :
  Diaphragmatic breathing,Segmental breathing, Incentive spirometer:
  Arms: Group A (Respiratory Training Group)
Other: Aerobic training — aerobic exercises are customized according to the patient's underlying disease and residual dysfunction. These exercises will include walking on treadmill. After an initial, 5-minute warm-up phase performed on the treadmill at a low load, each endurance training session lasted 30 minutes and ended with 5-minute recovery and relaxation phase. A total of 3-5 sessions are carried out per week. Patients who are prone to fatigue should perform intermittent exercises
  Arms: Group B : (Aerobic Training Group)

SUMMARY:
This study will be conducted on eighty patients of both sexes with age ranging from 35 to 45years. The will be recovered from COVID-19 infection with chest symptoms. They will be selected from Nasr city police authority hospital. They will be randomly assigned into 3 equal groups.

DETAILED DESCRIPTION:
This study will be conducted on eighty patients of both sexes with age ranging from 35 to 45years. The will be recovered from COVID-19 infection with chest symptoms. They will be selected from Nasr city police authority hospital. They will be randomly assigned into 3 equal groups.

Participants will be assigned into 3 groups equal in number (group A, group B, group C)

Group A (Respiratory Training Group) : It will include 30 patients of both sexes, recovered from COVID-19 infection. In addition to medical drugs, they will receive respiratory training for 6 weeks.

Group B : (Aerobic Training Group) : It will include 30 patients of both sexes, recovered from COVID-19 infection. In addition to medical drugs, they will receive aerobic training for 6 weeks

Group C : (control group) :It will include 20 patients of both sexes, recovered from COVID-19 infection on medical drugs only will receive no exercise as control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients recovered from COVID -19 infection.
* Patients with body mass index 25 - 35 kg/m2
* Patients previously diagnosed with chest symptoms of COVID- 19 infection.
* Patients' body temperature less than 37.5
* Blood oxygen saturation ≥95%

Exclusion Criteria:

* Smokers
* Patients with Myocardial infarction
* Patients with diabetes.
* Patients with autoimmune disease.
* Patients with positive COVID -19 infection.
* Patients with previous chest diseases
* a heart rate of >100 bpm
* a blood pressure of <90/60 mmHg or >140/90 mmHg
* a blood oxygen saturation of ≤95%
* other diseases that are not suitable for exercise (osteoarthritis knee - stroke patients, etc)

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Complete blood picture | change from baseline at 6 weeks
  A venous blood sample will be taken to be analyzed in the laboratory
Arterial blood gases | change from baseline at 6 weeks
  arterial blood sample will be assessed
6-minute walk Distance | change from baseline at 6 weeks
  patient will be instructed to walk as fast as long as possible, in a 30 meters obstacle- free corridor, limited by turnaround cones. Standardized verbal encouragement will be given every minute. After 6 min, patient will be instructed to stop, and the total distance will be measured, rounding to the nearest meter.
Breath-hold test | change from baseline at 6 weeks
  A rough index of cardiopulmonary reserve measured by the length of time that a person can voluntarily stop breathing; normal duration is 30 seconds or longer; diminished cardiac or pulmonary reserve is indicated by a duration of 20 seconds or less.
Oxygen saturation | change from baseline at 6 weeks
  Percentage of haemoglobin saturated with oxygen measured by pulse oximeter
Borg Dyspnea Scale score | change from baseline at 6 weeks
  It is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during six minute walk test

SECONDARY OUTCOMES:
Maximum oxygen consumption | change from baseline at 6 weeks
  Maximum oxygen consumption(VO2 max): Results of (6MWT) was used to calculate Vo2 max by using Cahalin equation as follows; Vo2 max = 0.03x distance in meters +3.98, in which distance is obtained from (6MWT)

CONTACTS AND LOCATIONS:
Locations (1):
- Police hospital-Nasr city, Cairo, Egypt